CLINICAL TRIAL: NCT07242651
Title: Effect of Tension and Trauma Releasing Exercises on Quality of Life and Sleep in Patients With Hypertension
Brief Title: Tension and Trauma Releasing Exercises on Hypertensive Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youmna Gamal Abdelmouty Elsayed, BSc. in Physical Therapy, Cairo University, 2018, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111995
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypertension (HTN)
Keywords: Tension and trauma releasing exercises
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study includes two parallel groups: the experimental group performs Tension and Trauma Releasing Exercises (TRE) in addition to medication, while the control group continues medication only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "TRE Exercise Group" (Experimental): Participants in this group will perform supervised Tension and Trauma Releasing Exercise (TRE) sessions in addition to their usual medical treatment for hypertension. The TRE sessions will be conducted three times per week for eight weeks, and each session will last approximately 30 minutes. The exercises aim to promote relaxation, reduce tension, and improve sleep quality, and quality of life.
  Interventions: Behavioral: Tension and trauma releasing exercises
- "Control Group" (No Intervention): Participants in this group will continue their usual medical treatment for hypertension without any additional exercise intervention. They will receive the same assessments for sleep quality, and quality of life as the experimental group.

INTERVENTIONS:
Behavioral: Tension and trauma releasing exercises — Tension and trauma releasing exercises will be conducted for study group only as follows: The exercises start by slightly fatiguing specific muscle groups to encourage this involuntary shaking, which is considered healthy and calming.
  The first exercise: Feet roll gently outward while shifting weight side to side, helping release ankle tension.
  The second exercise: One foot steps back while the front heel lifts until the calf feels lightly tired, triggering a small shake.
  The third exercise: A small lunge-like position engages the thighs and hips, leading to natural muscle release.
  The fourth exercise: A soft bend at the hips with relaxed arms and deep breathing stretches the back and encourages loosening.
  The fifth exercise: With feet wide and hands on the lower back, the hips push forward slightly while breathing deeply and turning gently side to side.
  The sixth exercise: The body slides into a seated position against a wall to lightly fatigue the
  Arms: "TRE Exercise Group"

SUMMARY:
The aim of this study is to investigate the effect of Tension and Trauma Releasing Exercises (TRE) on the quality of life and sleep in hypertensive patients. Participants will perform a series of supervised TRE sessions, and their sleep quality, and quality of life will be assessed before and after the intervention to determine any potential improvements related to the exercise.

DETAILED DESCRIPTION:
Forty females have had essential hypertension for at least five years. They will be recruited from the outpatient clinic at physical therapy, Cairo university.

The patients of this study will be randomly assigned into 2 equal groups (n=40):

Study Group A: (20 patients) Will receive Tension and Trauma Releasing Exercises in addition to medical treatment programme.

Control Group B: (20 patients) will receive only the Medical treatment programme.

The program of treatment for the study group will be applied 30 minutes per session , with a maximum of 15 minutes of neurogenic tremors, 3 times per week for 8 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be between 50 and 65 years of age.
2. The BMI of patients will range between 30 and 34.9.
3. Patients included in the study were diagnosed with essential hypertension for at least five years.
4. The patients will be in stage 1 hypertension under medical control, characterized by systolic blood pressure ranging from 140 to 159 mmHg and diastolic blood pressure ranging from 90 to 99 mmHg.

Exclusion Criteria:

1. Patients suffering from any unstable cardiovascular condition, such as uncontrolled arrhythmias or recent myocardial infarction.
2. Patients are diagnosed with secondary hypertension.
3. Patients with cognitive or physical impairments that prevent them from following instructions.

e) Patients who are taking beta-blockers and alpha-blockers because these medications may affect heart rate.

f) Individuals with endocrine disorders or any condition known to influence hormonal levels.

g) Patients are smokers. h) Malignant hypertension.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biological females only
Enrollment: 40 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Quality of life ,assessed by SF12 | Baseline and after 8 weeks of intervention
  Change in SF-12 physical and mental component summary scores from baseline to 8 weeks.
Sleep quality, assessed by the Pittsburgh Sleep Quality Index (PSQI). | Baseline and 8 weeks after the start of the intervention
  Change in global PSQI score from baseline to 8 weeks. PSQI will be administered to assess sleep quality .

SECONDARY OUTCOMES:
Blood pressure - Systolic and Diastolic (mmHg) ,assessed by mercury sphygmomanometer | Baseline and 8 weeks after the start of the intervention
  Mean change in systolic and diastolic blood pressure. Measurements will be taken using a mercury sphygmomanometer after a 5-minute rest period, and the average of two consecutive readings will be recorded.
Heart rate ,assessed by pulse oximeter | Baseline and 8 weeks after the start of the intervention
  change in resting heart rate measured by pulse oximeter
Depression and anxiety ,assessed by Hospital Anxiety and Depression Scale (HADS) | Baseline and 8 weeks after the start of the intervention
  Change in subscale (anxiety and depression) scores from baseline to 8 weeks.
Rate Pressure Product measurement | Baseline and 8 weeks after the start of the intervention
  Heart rate * systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: El-Sayed Essam Felaya, Assistant professor, Study Chair — Cairo University; Salma Elsayed Elsheikh, Lecturer of physical therapy, Study Chair — Cairo University; Mahmoud Mohamed Ghanema, Lecturer of Internal Medicine, Study Chair — Cairo University
Locations (1):
- Faculty of physical therapy ,Cairo University, Giza, Egypt